CLINICAL TRIAL: NCT03645720
Title: A Prospective Study of the Prognosis of Graft With Plastic Cannula in Hemodialysis
Brief Title: The Prognosis of Graft Using Plastic Cannula in Hemodialysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in performing study
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, choi sun ryoung, MD, Assistant professor, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-05-030
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal needle gruop (No Intervention): puncture using metal needle
- plastic cannula (Experimental): puncture using plastic cannula
  Interventions: Device: Plastic cannula

INTERVENTIONS:
Device: Plastic cannula — puncture using plastic cannula
  Arms: plastic cannula

SUMMARY:
The purpose of this study is to evaluate the complication of the puncture related complication in AVG (arteriovenous graft) such as pseudoaneurysm and hematoma, and the dialysis adequacy using plastic cannula versus metal needle in hemodialysis patients

DETAILED DESCRIPTION:
1. Ultrasonography is performed to determine the maturity of vascular access 4 weeks after AVG creation.
2. The first puncture is performed with plastic cannula or metal needle when it is judged that the blood vessel has matured.
3. Four skilled nurses perform vascular access puncture with plastic or metal needle
4. Ultrasound are used to evaluate and record the complications related to the puncture in plastic or metal needle group every month.
5. Complications and dialysis adequacy between the two groups will be evaluated after 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving hemodialysis treatment using AVG

Exclusion Criteria:

* Age under 20 years old or over 75 years old
* Abnormal skin condition using immunosuppressants such as steroids.
* Skin disorder
* Metal allergy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of pseudoaneurysm | Incidence of pseudoaneurysm at 6 months
  critical puncture related complication in AVG

SECONDARY OUTCOMES:
punctutre related complication | Monthly for 6 months.
  hematoma, inflitration, thrombus
Dialysis adeqaucy | Monthly for 6 months.
  Kt/V by serum test in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Sun Ryoung Choi, MD,PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No